CLINICAL TRIAL: NCT04841135
Title: Analysis of the Blood Signature of the Microbiota as a Diagnostic Marker of Alzheimer's Disease in the Early Stages of the Process: Pilot Study
Brief Title: Blood Microbiota Signature of Alzheimer's Disease
Acronym: MICMALZ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL19_0041
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Alzheimer Disease; Elderly With Normal Cognition
Keywords: Alzheimer; Memory; Aging; Microbiota
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alzheimer disease group (Other)
  Interventions: Other: Multiomics quantification; Other: Polysomnography
- Control (Other)
  Interventions: Other: Multiomics quantification; Other: Polysomnography
- Neurotypicals (Other)
  Interventions: Other: Multiomics quantification

INTERVENTIONS:
Other: Multiomics quantification — One time blood, stool and urine samples will be taken.
Other: Polysomnography — Facultative polysomnography
  Arms: Alzheimer disease group; Control

SUMMARY:
This study aims to validate a difference in blood microbial signature between Alzheimer's patients and control subjects in order to propose potential innovative strategies

DETAILED DESCRIPTION:
This is a pilot study only carried out in Montpellier, aimed at comparing AD patients with control subjects, including men / women aged between 50 and 85 years. The diagnosis of AD patients is based on international criteria. Metagenomics and proteomics will be used to determine the composition of the microbiota in whole blood and stools, but also the metabolomic profile in plasma, stool and the urines.

ELIGIBILITY:
Inclusion Criteria:

General criteria for AD and control groups:

* Male and/or female;
* Age between 50-85 years;
* Having given their free, informed, written consent, signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research);
* Patient benefiting from a social security scheme

AD group:

* Diagnosis of Alzheimer's disease according to the international ATN criteria of Albert et al, (1) who had a diagnostic lumbar puncture and CSF biomarker assay and brain imaging with analysis of hippocampal atrophy; topographic and pathophysiological markers must be positive to confirm the etiopathogenic diagnosis;
* Mild to moderate stage with MMSE score between 10 and 26 ;
* Symptomatic treatments specific to Alzheimer's disease (acetylcholinesterase inhibitors and memantine) and psychotropic treatments (anxiolytics, antidepressants, neuroleptics) are authorized but must be at fixed doses for more than 3 months ;

Control group:

- Patients seen in memory consultation for concern of having AD but for whom the workup is normal. These patients will have had a diagnostic lumbar puncture during the same memory consultation.

Neurotypical group criteria:

* Male and/or female ;
* Age between 18-35 years or between 50-85 years;
* Having given their free, informed, written and signed consent by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research);
* Patients without cognitive complaints seen in memory consultation but for whom the assessment is normal or young subjects recruited by advertisement. These participants will have an ex-post determination of plasma Aß and tau biomarkers.

Exclusion criteria:

General criteria for AD and control groups:

* Absence of a family caregiver to complete the neuropsychological scales and questionnaires ;
* Patient living in a medical institution;
* Illiteracy or inability to complete the psycho-behavioral tests;
* Major physical or neurosensory problems likely to interfere with the tests;
* Contra-indication or refusal to perform the biological tests;
* Refusal to carry out neuropsychological tests.
* Refusal of stool collection
* Digestive neoplasia in progress or < 5 years old
* Digestive surgery with intestinal resection ;
* Presence of inflammatory bowel disease or other familial gastrointestinal pathology ;
* Chronic use of laxatives;
* Antibiotics taken within one month prior to inclusion;
* Short-term life-threatening conditions (active cancer, unstable heart failure, severe liver, kidney and respiratory failure);
* Chronic psychosis or psychotic episodes;
* Alcohol or drug addiction;
* Epilepsy and other non-degenerative diseases of the central nervous system
* Vitamin B12 deficiency and unsupplemented folic acid ;
* Untreated hypothyroidism;
* Patient deprived of liberty, by judicial or administrative decision;
* Major protected by law;
* Patient in a period of relative exclusion from another protocol;
* Refusal to participate in the protocol.

AD group :

* Insufficient clinical and paraclinical information for the diagnosis of AD;
* Genetic form of AD (known genetic mutation);

Control and neurotypical groups: No specific non-inclusion criteria

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of bacterial 16S rDNA in stools | 22 months
  Concentration of bacterial 16S rDNA in stools

SECONDARY OUTCOMES:
Concentration of bacterial 16s DNA in blood | 22 months
  Concentration of bacterial 16s DNA in blood
Multiomics microbiota signature in AD | 22 months
  Multiomics microbiota signature in AD

CONTACTS AND LOCATIONS:
Overall Officials: Karim BENNYS, MD, PhD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier university hospital, Montpellier, France